CLINICAL TRIAL: NCT05882825
Title: The Level of Knowledge and Awareness of Dry Needling Treatment in the Turkish Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: DNK1
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Dry Needling

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to the physical medicine and rehabilitation outpatient clinic.: Patients admitted to the physical medicine and rehabilitation outpatient clinic and gave consent to participate.
  Interventions: Other: Dry Needling Therapy Knowledge and Awareness Questionnaire

INTERVENTIONS:
Other: Dry Needling Therapy Knowledge and Awareness Questionnaire — Dry Needling Therapy Knowledge and Awareness Questionnaire is a questionnaire consisting of a total of 14 questions created by the researchers who are specialized in the field. The correct answer to each question is one point. A high score indicates a high level of knowledge and awareness, while a low score indicates a low level of awareness and knowledge.

SUMMARY:
The study will employ a cross-sectional design to assess the level of knowledge and awareness of dry needling therapy in the Turkish population.

DETAILED DESCRIPTION:
A representative sample of individuals will be selected for participation in the survey. A structured questionnaire will be developed specifically for this study, consisting of questions related to the knowledge and awareness of dry needling therapy. The questionnaire will be administered through face-to-face interviews. Data collected from the survey will be analyzed using appropriate statistical methods to determine the overall level of knowledge and awareness of dry needling therapy among the Turkish population.

ELIGIBILITY:
Inclusion Criteria:

* Giving consent.

Exclusion Criteria:

* Not giving consent.
* Any illness or disability that can prevent filling out the form or communicating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to the physical medicine and rehabilitation outpatient clinic and gave consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Level of Knowledge and Awareness of Dry Needling Therapy in the Turkish Population | 1 day
  By using the data gained with the Dry Needling Therapy Knowledge and Awareness Questionnaire and using the suggested statistical methods by the statistics expert, this study will aim to determine the level of knowledge and awareness of myofascial pain syndrome in the Turkish population.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data will be shared upon reasonable request by the corresponding author.